CLINICAL TRIAL: NCT07155356
Title: Effect of Red and Blue Light Irradiation on Postoperative Wound Healing in Perianal Abscess: a Single-center Prospective Open-label Randomized Clinical Trial
Brief Title: Effect of Red and Blue Light Irradiation on Postoperative Wound Healing in Perianal Absces
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHPutianU-012
Record Dates: First submitted 2025-07-31; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Perianal Abscess
Keywords: perianal abscess; red light phototherapy; red and blue light phototherapy; wound healing
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Routine care of patients after surgery for perianal abscesses.
- Red Ligh Group (Experimental): Postoperative care of patients with perianal abscesses using routine plus red light irradiation.
  Interventions: Device: Red light exposure
- Combined Red-Blue Light Group (Experimental): Use of routine plus red and blue light in postoperative care of patients with perianal abscesses.
  Interventions: Device: Red-blue light exposure

INTERVENTIONS:
Device: Red light exposure — Patients in the red light group received red light therapy concurrently with standard care.
  Arms: Red Ligh Group
Device: Red-blue light exposure — Patients in the red and blue light group received combined red and blue light therapy concurrently with standard care。
  Arms: Combined Red-Blue Light Group

SUMMARY:
This study aims to investigate whether specialized red-blue light irradiation facilitates faster postoperative recovery and reduces complication rates in patients following perianal abscess surgery. A total of 222 eligible patients were randomly allocated equally into three groups (74 per group):①Routine Care Group: Standard wound care including cleansing and dressing changes；②Red Light Therapy Group: Routine care plus red light phototherapy；③Combined Red-Blue Light Therapy Group: Routine care plus concurrent red and blue light phototherapy.Wound healing time and incidence of complications were compared to assess postoperative recovery across interventions. The primary hypothesis posits that adjunctive phototherapy-particularly combined red-blue light irradiation-will significantly enhance wound healing, reduce edema and pain, and decrease complication rates (e.g.bleeding, urinary retention) compared to routine care alone.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years;
* Clinical diagnosis of perianal abscess；
* Procedure: Radical resection with incision and drainage.

Exclusion Criteria:

* Concurrent anorectal disorders (hemorrhoids, anal fissure) or malignancies/infectious diseases；
* History of psychiatric disorders；
* Analgesic use within 7 days preoperatively；
* Coagulopathy or cardiac/hepatic dysfunction；
* Pregnancy or lactation；
* Contraindications to phototherapy；
* IBD-related perianal abscess.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-08-14 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | Measurements were taken over a time frame of 24 hours postoperatively to complete epithelialisation.
  Defined as 100% re-epithelialization assessed by blinded evaluator.

SECONDARY OUTCOMES:
Postoperative pain intensity | Baseline, Day 1, 3, 5, 7, and Day 14±2
  Assessed at rest and during defecation.Numerical Rating Scale will be used,patients are asked to choose a whole number (integer) from 0 to 10 that best describes their pain.0 usually means "no pain."10 means "the worst pain imaginable."
Peripheral tissue edema（Grade 0-3） | Day 1, 3, 5, 7, and Day 14±2
  * Grade 0 (None): No edema.
  * Grade 1 (Mild): Mild edema with slight swelling around the incision; skin folds remain clearly visible.
  * Grade 2 (Moderate): Moderate edema with pronounced swelling around the incision; skin folds are indistinct.
  * Grade 3 (Severe): Severe edema with marked swelling around the incision; skin folds are obliterated.
Assessment of Granulation Tissue in Wound Bed | Day 1, 3, 5, 7, and Day 14±2
  * Grade 0 (Absent): No granulation tissue present.
  * Grade 1 (Poor): Minimal, pale, and friable granulation tissue with easy bleeding.
  * Grade 2 (Fair): Moderate amount of granulation tissue; pinkish-red in color but remains somewhat friable.
  * Grade 3 (Good): Healthy, abundant granulation tissue filling the wound bed; beefy red in color and firm to the touch, with minimal bleeding.
Length of hospital stay | From surgery end to discharge (up to 7 days)
  Measured in hours with standardized discharge criteria.
Complication incidence | Within 30 days postoperatively
  Measurements include the incidence of postoperative bleeding, urinary retention, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Putian University, Putian, China

IPD SHARING:
Plan to Share IPD: No
Based on a strict commitment to participant privacy protection, compliance with the terms of the ethical review protocol, and adherence to the sponsoring institution's policies, IPD from this study will not be shared at this time.